CLINICAL TRIAL: NCT05271643
Title: Preventing Depression and Anxiety: a Pilot Study of a Cystic-fibrosis Specific Cognitive-behavioral Therapy Intervention for Adolescents With CF
Brief Title: Pilot Study of a CF-specific CBT Intervention for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University at Buffalo (Other); University of Kansas Medical Center (Other); Behavioral Health Systems Research (Unknown)
Responsible Party: Principal Investigator, Deborah Friedman, Assistant Professor of Psychology (Psychiatry), Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P001492
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis; Depression; Anxiety
MeSH Terms: conditions — Cystic Fibrosis; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CF-CBT-A intervention (Experimental): Participants will meet with a therapist, a mental health provider on their cystic fibrosis care team who has received training in CF-CBT-A, for a baseline interview and introduction plus 9 weekly sessions of CF-CBT-A.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — CF-CBT-A is an 10-session program for adolescents with cystic fibrosis introducing cognitive-behavioral coping skills for managing stress, and for prevention and treatment of anxiety and depression. The content of the program was developed to address stressors related to coping with cystic fibrosis. Participants will receive a patient workbook, and meet with a trained mental health clinician on their CF team who will guide them through learning and practicing coping skills. Parents/guardians involvement will be encouraged. A parent/guardian will attend the baseline and final session, have the opportunity for a mid-program check-in, and receive a workbook of psychoeducational material that parallels the adolescent workbook, featuring tips for supporting their teens, and weekly e-mail communication.

SUMMARY:
The goal of this study is to pilot a new CF-specific cognitive-behavioral therapy intervention (CF-CBT-A) for prevention and treatment of depression and anxiety for adolescents with CF. CF-CBT-A is a 10-session program that was developed with input from adolescents with CF and parents and CF care teams to be highly relevant to the unique needs of adolescents with CF. The program will be piloted at 3 U.S. CF centers with 10 to 12 adolescents with cystic fibrosis who have mild to moderately severe symptoms of depression and/or mild to severe symptoms of anxiety. It will be delivered by mental health coordinator members of the participant's CF care team who receive training, with sessions occurring in-person or via telehealth. We will examine feasibility and acceptability of the intervention as indicated by measures of completion, intervention fidelity, and adolescent and parent satisfaction ratings. We will also examine preliminary evidence of effectiveness. If this intervention is successful, symptoms of depression and anxiety and perceived psychological stress will decrease and coping self-efficacy and health-related quality of life (HRQoL) will improve.

ELIGIBILITY:
Inclusion Criteria:

1. Be 12-17 years of age
2. Have a diagnosis of CF
3. 3. Have depression symptom scores on the PHQ-A in the mild to moderately severe range (> 4 and ≤ 19), but not in the severe range, and/or anxiety scores on the GAD-7 from mild to severe range (5 to 21).
4. Be able to speak and read English
5. Be willing and able to provide assent
6. Have a parent who is willing and able to provide informed consent for their own and adolescent participation
7. Have a parent who is able to speak and read English; the parent will participate in the study in support of their adolescent during the intervention and complete pre- and post- assessments.
8. Subjects will not be excluded for the following reasons:

   1. CF severity or lung/liver transplant status, if they are otherwise able to participate in CBT. If subjects are medically hospitalized during the course of the study, they may continue to participate in the CBT intervention or follow up visits during or following hospitalization as clinically appropriate.
   2. A history of more severe depression currently at mild to moderate levels with or without treatment.
   3. Participation in concomitant psychosocial treatments (with the exception of formal CBT) or psychopharmacologic treatments at baseline, although these concomitant treatments will be tracked and considered in analysis.

Exclusion criteria:

1. Any subjects who are deemed to present an acute safety risk to self or others will be excluded. Subjects reporting a positive answer on question 9 on the PHQ-9, dealing with suicidality, will be further assessed for severity and clinical context, including administration of the Columbia Suicide Severity Rating Scale (C-SSRS, Screen Version, Recent; Posner, 2011). Those reporting suicidal intent with or without specific plan (yes to question 4 and/or 5 on the C-SSRS) will be excluded from the study. These individuals will be referred for urgent/emergent further assessment and treatment as clinically indicated.

2) Participation in concomitant formal cognitive-behavioral therapy at baseline

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Treatment acceptability as measured by item and total score summation on the Client Satisfaction Questionnaire (CSQ-8) with additional study-specific items | immediately post-intervention
  TThe Client Satisfaction Questionnaire (CSQ-8) is an 8-item self-report measure that assesses patient service satisfaction,rated on a 4-point scale from 1=lowest to 4=highest satisfaction. Post-intervention treatment satisfaction will also be assessed with a series of structured and open-ended questions specific to the study intervention. Completed by parent and adolescent. Assessed one time immediately post-intervention.
Feasibility of the intervention will be indicated by Rate of completion of the CF-CBT-A program sessions once enrolled | From baseline to post-intervention (2-3 months)
  Rate of complete will be summarized by calculating the percentage of CF-CBT-A sessions completed by participants over the course of the study period.

SECONDARY OUTCOMES:
Change from baseline in Depressive symptoms measured by the Patient Health Questionnaire-9 (PHQ-9) - adolescent version | From baseline to post-intervention (2-3 months)
  The PHQ-9 consists of nine questions measuring frequency of depressive symptoms, rated on a Likert scale from 0 "not at all" to 3 "nearly every day," with total score ranging 0-27. Clinical severity scores have been established with scores of 5, 10, 15, and 20 representing cut-off scores for mild, moderate, moderately severe, and severe depression, respectively.
Change from baseline in Anxiety symptoms measured by the Generalized Anxiety Disorder-7 item scale (GAD-7) | From baseline to post-intervention (2-3 months)
  The GAD-7 is a 7-item measure of symptoms of anxiety. Likert scale ratings allow total scores of 0-21. Scores of 5, 10, and 15 correspond to severity ratings of mild, moderate and severe anxiety.
Change in Perceived Stress, measured by the PROMIS Pediatric and Parent Proxy Psychological Stress Experiences 8-item short forms | From baseline to post-intervention (2-3 months)
  This measure assesses psychological stress reactions (e.g., feeling overwhelmed, perceived lack of control of capacity to manage one's life).5Adolescents will self-report and parents will complete the proxy report about their child, providing another perspective on adolescent adjustment. Both scales use a 7-day recall period and include 8 items rated on a 5-point Likert Scale from "Never" to "Always," (e.g., In the past 7 days, I felt stressed).
Change in Health-Related Quality of Life, measured by the Cystic Fibrosis Questionnaire-Revised (CFQ-R) | From baseline to post-intervention (2-3 months)
  The CFQ-R is a well-established measure of HRQoL, validated in a national, multicenter longitudinal study, and demonstrating consistent associations with health outcomes. A parent proxy version will be administered for adolescent participants ages 12 and 13.
Change in Coping Self-Efficacy, measured by the CF Coping Self-Efficacy Scale - adolescent version | From baseline to post-intervention (2-3 months)
  A self-report measure of confidence in being able to cope with the daily challenges associated with CF developed with input of people with CF. Confidence in being able to use coping skills targeted by the intervention, including those specific to coping with CF, are rated on a 10-point scale from 'very sure' to 'very unsure'.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Friedman, PhD, Principal Investigator — Massachusetts General Hospital (MGH); Anna M Georgiopoulos, MD, Principal Investigator — Massachusetts General Hospital (MGH)
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University at Buffalo, New York, New York

IPD SHARING:
Plan to Share IPD: No